CLINICAL TRIAL: NCT02176915
Title: Fresh Start: A Randomized Clinical Trial
Brief Title: Trial of Fresh Start Weight Loss Intervention in WIC Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Stephenie Lemon, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1P60MD006912 (NIH); P60MD006912 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group program (Experimental): 8-session group weight loss program and 4 follow-up phone counseling sessions
  Interventions: Behavioral: Group program
- Print Materials (Active Comparator): 8 weekly mailings of print materials covering weight loss topics through US mail.
  Interventions: Behavioral: Print Materials

INTERVENTIONS:
Behavioral: Group program
  Arms: Group program
Behavioral: Print Materials
  Arms: Print Materials

SUMMARY:
The Fresh Start postpartum weight loss program will test the effectiveness of a group-based weight loss intervention that includes videos featuring peers who have successfully achieved postpartum weight loss. The group-based condition will be compared to a control condition involving print materials related to weight loss.

DETAILED DESCRIPTION:
The goal is to study the effectiveness and implementation of a postpartum weight loss intervention for WIC clients that has potential for sustainability. The investigators will compare outcomes among participants in a group-based weight loss intervention condition (Fresh Start) to outcomes among participants in a self-directed, print materials only, comparison group. The Fresh Start intervention, informed by formative research studies, consists of an 8-session group-based weight loss intervention delivered by WIC nutritionists and peer leaders. The intervention integrates key educational and skill building strategies from the lifestyle arm of the Diabetes Prevention Program with delivery strategies and messages specific for the WIC program and postpartum women. The intervention will be evaluated in a randomized clinical trial that will contribute to generalizable knowledge.

ELIGIBILITY:
Inclusion Criteria:

* 6 months or less postpartum
* Speaks English
* BMI 25 or greater
* Client of WIC program, Worcester MA

Exclusion Criteria:

* Not able to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-07; Primary Completion 2018-12 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index from baseline | 3 months, 12 months

SECONDARY OUTCOMES:
Change in Pregnancy Physical Activity Questionnaire score from baseline | 3 months, 12 months
Change in 24-hour dietary recall from baseline | 3 months, 12 months
  Dietary behavior will be measured using a 24-hour dietary recall.

CONTACTS AND LOCATIONS:
Overall Officials: Stephenie Lemon, PhD, Principal Investigator — UMass Worcester
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Rosal MC, Haughton CF, Estabrook BB, Wang ML, Chiriboga G, Nguyen OH, Person SD, Lemon SC. Fresh Start, a postpartum weight loss intervention for diverse low-income women: design and methods for a randomized clinical trial. BMC Public Health. 2016 Sep 9;16(1):953. doi: 10.1186/s12889-016-3520-0. PMID 27612615